CLINICAL TRIAL: NCT00001149
Title: Monitoring of Seizures, EEG and Serum Antiepileptic Drug Concentrations in Patients With Uncontrolled Epilepsy
Brief Title: Monitoring Patients With Uncontrolled Epilepsy
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 750124; 75-N-0124
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-01

CONDITIONS: Epilepsy; Seizures
Keywords: Anticonvulsants; Intensive Monitoring; Epilepsy
MeSH Terms: conditions — Epilepsy; Seizures

SUMMARY:
This study is designed to evaluate patients with uncontrolled seizures. Seizures can be associated with and monitored by abnormal electrical activity in the brain.

In this study researchers will use video-electroencephalography (EEG) to monitor patients with uncontrolled or suspected seizures. EEG works by measuring electrical activity in different areas of the brain. The video-EEG allows researchers to examine changes in the EEG along with the clinical features of seizures as they occur.

In addition to monitoring electrical activity of the brain, researchers will take frequent antiepileptic drug blood levels. These measures will allow researchers to learn more about how each drug is absorbed and metabolized in the body.

The information collected in the study will be used to place patients into other scientific studies testing new therapies for epilepsy.

DETAILED DESCRIPTION:
In this study we will use standard clinical studies, including simultaneous Video-EEG monitoring, to evaluate patients referred for uncontrolled or suspected seizures. The protocol will be used to screen patients for inclusion in other protocols, follow the natural history of seizure disorders, and train fellows in the evaluation and treatment of epilepsy. Both inpatients and outpatients will be studied.

ELIGIBILITY:
History of uncontrolled seizures, at the present time, at least during 6 months of the past 3 years, and preferably a continuous pattern of seizures during the few months prior to admission.

Seizure frequency, by history, must be sufficient to make video monitoring effective. Priority will be given to patients whose seizures occur once or more per day.

Patients of any age may be accepted.

Patients (and parents or guardians, if applicable) must express willingness to cooperate with the entire protocol, to be willing to undergo further diagnostic tests if needed, and to return for follow up evaluation at intervals as needed.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 900
Dates: Start 1975-11; Study Completion 2002-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Theodore WH, Porter RJ, Penry JK. Complex partial seizures: clinical characteristics and differential diagnosis. Neurology. 1983 Sep;33(9):1115-21. doi: 10.1212/wnl.33.9.11515. PMID 6684245
- [Background] Penry JK, Porter RJ, Dreifuss RE. Simultaneous recording of absence seizures with video tape and electroencephalography. A study of 374 seizures in 48 patients. Brain. 1975 Sep;98(3):427-40. doi: 10.1093/brain/98.3.427. PMID 1182486
- [Background] Altshuler LL, Devinsky O, Post RM, Theodore W. Depression, anxiety, and temporal lobe epilepsy. Laterality of focus and symptoms. Arch Neurol. 1990 Mar;47(3):284-8. doi: 10.1001/archneur.1990.00530030050016. PMID 2106868